CLINICAL TRIAL: NCT02900378
Title: A Multi-center, Prospective, Randomized, Double-blind Study to Assess the Impact of Sacubitril/Valsartan vs. Enalapril on Daily Physical Activity Using a Wrist Worn Actigraphy Device in Adult Chronic Heart Failure Patients
Brief Title: randOmized stUdy Using acceleromeTry to Compare Sacubitril/valsarTan and Enalapril in Patients With Heart Failure
Acronym: OUTSTEP-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLCZ696B3301; 2016-003085-32 (EudraCT Number)
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction
Keywords: sacubitril/valsartan; enalapril; physical activity; actigraphy; sleep; heart failure; reduced ejection fraction; randomized controlled trial; accelerometry
MeSH Terms: conditions — Motor Activity; Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; sacubitril; Valsartan; Enalapril

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LCZ696 (Sacubitril/Valsartan) (Experimental): After randomization, patients in this arm received LCZ696 (Sacubitril/Valsartan) twice daily and matching placebo of Enalapril depending on the patient's previous ACEI/ARB dose (enalapril equivalent dose) for 2 weeks. Patients could start study medication at dose level 1 (24 mg/26 mg LCZ), 2 (49 mg/51 mg LCZ) or 2a (49 mg/51 mg LCZ) or matching placebo bid. After 2 weeks (visit 3) the doses were up-titrated: patients, who started on dose level 2 or 2a received the target dose of study medication (level 3) at this point. After another 2 weeks (visit 4) all patients were to achieve the target dose of 97 mg/103 mg bid LCZ696(sacubitril/valsartan) and matching placebo, provided no safety and tolerability issues arised during uptitration.
  Interventions: Drug: LCZ696 (Sacubitril/Valsartan); Drug: Placebo of Enalapril
- Enalapril (Active Comparator): After randomization, patients in this arm received Enalapril twice daily and matching placebo of LCZ696 (Sacubitril/Valsartan) depending on the patient's previous ACEI/ARB for 2 weeks. Patients could start study medication at dose level 1 or 2a or matching placebo bid. After 2 weeks (visit 3) the doses were up-titrated: patients, who started on dose level 2 or 2a received the target dose of study medication (level 3) at this point. After another 2 weeks (visit 4) all patients were to achieve the target dose of 10 mg bid enalapril and matching placebo, provided no safety and tolerability issues arised during uptitration
  Interventions: Drug: Placebo of LCZ696 (Sacubitril/Valsartan); Drug: Enalapril

INTERVENTIONS:
Drug: LCZ696 (Sacubitril/Valsartan) — LCZ696 (sacubitril/valsartan) was available in 24 mg/26 mg, 49 mg/51 and 97 mg/103 mg mg film-coated tablets
  Other Names: LCZ696
  Arms: LCZ696 (Sacubitril/Valsartan)
Drug: Placebo of LCZ696 (Sacubitril/Valsartan) — Placebo of LCZ696 (sacubitril/valsartan) was available to match 24 mg/26 mg, 49 mg/51 and 97 mg/103 mg mg film-coated tablets
  Other Names: Placebo
  Arms: Enalapril
Drug: Enalapril — Enalapril was available in 2.5 mg, 5 mg and 10 mg film-coated tablets
  Arms: Enalapril
Drug: Placebo of Enalapril — Placebo of Enalapril was available to match 2.5 mg, 5 mg and 10 mg film-coated tablets
  Other Names: Placebo
  Arms: LCZ696 (Sacubitril/Valsartan)

SUMMARY:
The purpose of this randomized, actively controlled, double-blind study with prospective data collection was to assess differences between sacubitril/valsartan versus enalapril in increasing exercise capacity and non-sedentary physical activity in HFrEF patients. Physical activity was assessed by the 6 minute walk test, and daily physical activity was continuously measured by means of a wrist-worn accelerometry device from 2 weeks before until 12 weeks after start of study therapy (sacubitril/valsartan or enalapril).

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent obtained before any study assessment is performed.
* Ambulatory ≥ 18 years of age with a diagnosis of chronic symptomatic HF (NYHA class ≥ II) with reduced ejection fraction, defined as known LVEF ≤ 40%

AND one of the following two criteria:

* Plasma NT-proBNP level of ≥ 300 pg/mL or BNP ≥ 100 pg/mL (measurement may be recorded no longer than past 12 months) OR
* Confirmation of a heart failure hospitalization last 12 months.
* Patients must be on stable HF medication for at least 4 weeks prior to Week - 2, where the minimal daily dose of current evidence based therapies is equivalent to at least 2.5 mg/d enalapril
* Willingness to wear the accelerometer wristband continuously for the duration of the trial.
* Patients must be living in a setting, allowing them to move about freely and where they are primarily self-responsible for scheduling their sleep and daily activities.

Key Exclusion Criteria:

* History of hypersensitivity to any of the study drugs or their excipients or to drugs of similar chemical classes
* Use of sacubitril/valsartan prior to week - 2.
* Bedridden patients, or patients with significantly impaired/limited physical activity and/or fatigue due to medical conditions other than HF, such as, but not limited to angina (chest pain at exertion), arthritis, gout, peripheral artery occlusive disease, obstructive or restrictive lung disease, malignant disease, neurological disorders (e.g. Parkinson's or Alzheimer's disease, central and peripheral neuroinflammatory and -degenerative disorders or functional central nervous lesions due to hemodynamic or traumatic incidents), injuries (incl. diabetic foot ulcers) or missing limbs
* Patients with palsy, tremor or rigor affecting the non-dominant arm.
* Patients with any skin or other condition of the non-dominant arm that would limit the ability to wear the actigraphy device continuously (24h/day) over 14 weeks.
* Patients fully depending on a mobility support system, e.g. wheelchair, scooter or walker. Patients are allowed to use a cane as long as this is not used with the non-dominant arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (106):
- Belgium (5):
  - Novartis Investigative Site, Edegem, Antwerpen
  - Novartis Investigative Site, Dendermonde
  - Novartis Investigative Site, Geel
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Turnhout
- Bulgaria (3):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
- Czechia (6):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Chomutov, Czech Republic
  - Novartis Investigative Site, Svitavy, Czech Republic
  - Novartis Investigative Site, Most, CZE
  - Novartis Investigative Site, Kolín
  - Novartis Investigative Site, Prague
- Denmark (5):
  - Novartis Investigative Site, Elsinore
  - Novartis Investigative Site, Odense C
  - Novartis Investigative Site, Randers
  - Novartis Investigative Site, Roskilde
  - Novartis Investigative Site, Svendborg
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Finland (2):
  - Novartis Investigative Site, Hämeenlinna
  - Novartis Investigative Site, Tampere
- France (3):
  - Novartis Investigative Site, Auxerre
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Metz-Tessy
- Germany (22):
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Bad Homburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Buchholz in der Nordheide
  - Novartis Investigative Site, Dietzenbach
  - Novartis Investigative Site, Elsterwerda
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Halberstadt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Haßloch
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Löhne
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Mühldorf
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Reinfeld
  - Novartis Investigative Site, Schwäbisch Hall
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Wallerfing
  - Novartis Investigative Site, Wedel
  - Novartis Investigative Site, Wermsdorf
- Greece (4):
  - Novartis Investigative Site, Alexandroupoli, Evros
  - Novartis Investigative Site, Heraklion Crete, Greece
  - Novartis Investigative Site, Voula, GR
  - Novartis Investigative Site, Athens
- Iceland (2):
  - Novartis Investigative Site, Kopavogur
  - Novartis Investigative Site, Reykjavik
- Novartis Investigative Site, Dublin, Ireland
- Latvia (3):
  - Novartis Investigative Site, Jelgava
  - Novartis Investigative Site, Ogre
  - Novartis Investigative Site, Riga
- Lithuania (3):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Klaipėda, LTU
  - Novartis Investigative Site, Vilnius
- Netherlands (6):
  - Novartis Investigative Site, Goes
  - Novartis Investigative Site, Haarlem
  - Novartis Investigative Site, Heerlen
  - Novartis Investigative Site, Leiderdorp
  - Novartis Investigative Site, Roermond
  - Novartis Investigative Site, Veldhoven
- Novartis Investigative Site, Feiring, Norway
- Poland (3):
  - Novartis Investigative Site, Warsaw, Masovian Voivodeship
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Lodz, Łódź Voivodeship
- Spain (24):
  - Novartis Investigative Site, Ferrol, A Coruna
  - Novartis Investigative Site, Elche, Alicante
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Huelva, Andalusia
  - Novartis Investigative Site, Sanlúcar de Barrameda, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Villamartín, Cadiz
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Aranda de Duero, Castille and León
  - Novartis Investigative Site, Burgos, Castille and León
  - Novartis Investigative Site, León, Castille and León
  - Novartis Investigative Site, Soria, Castille and León
  - Novartis Investigative Site, Sabadell, Catalonia
  - Novartis Investigative Site, Cáceres, Extremadura
  - Novartis Investigative Site, Lugo, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Gijón, Principality of Asturias
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Manises, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Girona
  - Novartis Investigative Site, Madrid
- Sweden (3):
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Mölndal
  - Novartis Investigative Site, Stockholm
- United Kingdom (8):
  - Novartis Investigative Site, Stockton-on-Tees, Cleveland
  - Novartis Investigative Site, Rothwell, GBR
  - Novartis Investigative Site, Faringdon, Oxfordshire
  - Novartis Investigative Site, Gateshead, Tyne and Wear
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, Cumbria
  - Novartis Investigative Site, Poole
  - Novartis Investigative Site, Wellingborough

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 120 centers in 19 countries worldwide (Belgium, Bulgaria, Czech Republic, Denmark, Estonia, Finland, France, Germany, Greece, Iceland, Ireland, Latvia, Lithuania, Netherlands, Norway, Poland, Spain, Sweden and UK).
Pre-assignment Details: It was planned to recruit 300 patients per treatment arm, i.e. 600 patients in total. A total of 764 patients were screened, of whom 621 patients were randomized (310 in the sacubitril/valsartan group and 311 in the enalapril group).
Groups:
- LCZ696 (Sacubitril/Valsartan): LCZ696 (Sacubitril/Valsartan) or its matching placebo twice a day for 12 weeks. Patients began study treatment (Sacubitril/Valsartan) at a specific dose level according to their pre-study ACEI/ARB dose (1 (24 mg/26 mg LCZ), 2 (49 mg/51 mg LCZ) or 2a (49 mg/51 mg LCZ)) or matching placebo and were up-titrated according to an up-titration scheme.
- Enalapril: Enalapril or its matching placebo twice a day for 12 weeks. Patients began study treatment (Enalapril) at a specific dose level according to their pre-study ACEI/ARB dose (1 (2.5 mg), 2a (5 mg)) or matching placebo and were up-titrated according to an up-titration scheme.
Period: Randomization (Visit 2)
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Started (All randomized patients) | 310 | 311
Completed | 287 | 283
Not Completed | 23 | 28
Not completed — Adverse Event | 14 | 11
Not completed — Death | 1 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Non-compliance with Study Drug | 1 | 1
Not completed — Protocol Deviation | 1 | 7
Not completed — Withdrawal by Parent/Guardian | 5 | 3
Not completed — Withdrawal of Informed Consent | 0 | 2
Period: Treatment Phase
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Started (All randomized patients with at least 1 dose of study treatment) | 309 | 310
Full Analysis Set (At least 1 dose of study treatment and 1 post baseline safety assessment) | 302 | 302
Completed | 309 | 310
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients are represented in the overall number of Baseline Participants. The Demographic and Baseline Characteristics were done in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril | Total
Number analyzed (Participants) | 310 | 311 | 621
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The Demographic and Baseline Characteristics were done in the Safety Analysis Set.
  Years
    number analyzed (Participants) | 309 | 310 | 619
    (all) | 67.16 (11.04) | 66.62 (10.45) | 66.89 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Demographic and Baseline Characteristics were done in the Safety Analysis Set.
  Participants
    number analyzed (Participants) | 309 | 310 | 619
    Female | 71 | 61 | 132
    Male | 238 | 249 | 487
Race/Ethnicity, Customized [Number; unit: Participants] — Population: The Demographic and Baseline Characteristics were done in the Safety Analysis Set.
  Participants
    Black or African American: number analyzed (Participants) | 309 | 310 | 619
    Black or African American | 1 | 0 | 1
    White: number analyzed (Participants) | 309 | 310 | 619
    White | 298 | 299 | 597
    Missing: number analyzed (Participants) | 309 | 310 | 619
    Missing | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Week 0) in the Six Minute Walk Test (6MWT) at End of Study (Week 12)
Description: The impact of LCZ696 (Sacubitril/Valsartan) and Enalapril on functional exercise capacity was measured by the Six Minute Walk Test at 12 weeks. The 6MWT measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is able to self-pace and rest as needed as they traverse back and forth along a marked walkway.
Time Frame: Baseline, Week 12
Population: The Full Analysis Set (FAS) and FAS population subset without AE/SAE were considered
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 302 | 302
meters
  Baseline (FAS): number analyzed (Participants) | 301 | 300
  Baseline (FAS) | 365.37 (108.18) | 371.08 (104.41)
  Week 12 (FAS): number analyzed (Participants) | 292 | 284
  Week 12 (FAS) | 395.80 (113.11) | 395.33 (105.94)
  Change from BL at Week 12 (FAS): number analyzed (Participants) | 291 | 282
  Change from BL at Week 12 (FAS) | 31.57 (67.35) | 24.89 (51.64)
  Baseline (FAS without AE/SAE): number analyzed (Participants) | 289 | 292
  Baseline (FAS without AE/SAE) | 364.72 (106.86) | 371.18 (105.13)
  Week 12 (FAS without AE/SAE): number analyzed (Participants) | 283 | 277
  Week 12 (FAS without AE/SAE) | 399.31 (110.54) | 396.02 (106.39)
  Change from BL at Week 12 (FAS without AE/SAE): number analyzed (Participants) | 282 | 275
  Change from BL at Week 12 (FAS without AE/SAE) | 35.75 (58.76) | 25.87 (51.73)
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 12 (FAS); Test type: Other; p = 0.2464, ANCOVA — The comparison of treatment groups were out using an analysis of covariance (ANCOVA) model adjusting for treatment and baseline NYHA class (NYHA II vs. III/IV) and the 6MWT baseline value as covariates; Differences of least square means = 5.68, 95% CI 2-sided [-3.93 to 15.29], Standard Error of Mean 4.89
Statistical Analysis 2: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 12 (FAS without AE/SAE); Test type: Other; p = 0.0503, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Differences of least square means = 8.98, 97.5% CI 2-sided [-1.31 to 19.27], Standard Error of Mean 4.58

2. Primary Outcome: Change From Baseline (Week 0) in Mean Daily Non-sedentary Daytime Activity at End of Study (Week 12)
Description: Non-sedentary physical activity is defined as >= 178.50 activity counts per minute; the average number of minutes per day spent in non-sedentary physical activity is being calculated over 14 days before randomization (baseline i.e. week -2 to week 0) and the last 14 days of treatment (i.e. week 10 to week 12).
Time Frame: Baseline, Week 12
Population: The FAS population with Multiple Imputation (MI), with Last Observation Carried Forward (LOCF) and without MI/LOCF were considered.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 302 | 302
minutes
  Baseline (FAS with MI) | 510.11 (128.08) | 506.81 (139.60)
  Week 12 (FAS with MI) | 479.69 (124.23) | 487.53 (126.84)
  Change from BL at Week 12 (FAS with MI) | -30.42 (102.55) | -19.28 (104.04)
  Baseline (FAS with LOCF): number analyzed (Participants) | 259 | 257
  Baseline (FAS with LOCF) | 512.07 (126.37) | 505.31 (129.74)
  Week 12 (FAS with LOCF): number analyzed (Participants) | 253 | 256
  Week 12 (FAS with LOCF) | 489.43 (127.36) | 490.09 (127.82)
  Change from BL at Week 12 (FAS with LOCF): number analyzed (Participants) | 253 | 256
  Change from BL at Week 12 (FAS with LOCF) | -21.88 (68.55) | -15.41 (74.45)
  Baseline (FAS without MI/LOCF): number analyzed (Participants) | 259 | 257
  Baseline (FAS without MI/LOCF) | 512.07 (126.37) | 505.31 (129.74)
  Week 12 (FAS without MI/LOCF): number analyzed (Participants) | 234 | 216
  Week 12 (FAS without MI/LOCF) | 479.81 (122.45) | 486.85 (128.70)
  Change from BL at Week 12 (FAS without MI/LOCF): number analyzed (Participants) | 203 | 194
  Change from BL at Week 12 (FAS without MI/LOCF) | -25.14 (69.11) | -20.51 (72.52)
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 12 (FAS with MI); Test type: Other; p = 0.4769, ANCOVA — The comparison of treatment groups were carried out using an ANCOVA model adjusting for treatment, baseline NYHA class (NYHA II vs. III/IV) and the daily non-sedentary daytime activity baseline value as covariates; Differences of least square means = -6.14, 97.5% CI 2-sided [-25.70 to 13.41], Standard Error of Mean 8.61
Statistical Analysis 2: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 12 (FAS with LOCF); Test type: Other; p = 0.3463, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Differences of least square means = -5.67, 95% CI 2-sided [-17.48 to 6.14], Standard Error of Mean 6.01
Statistical Analysis 3: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 12 (FAS without MI/LOCF); Test type: Other; p = 0.3513, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Differences of least square means = -6.24, 95% CI 2-sided [-19.39 to 6.91], Standard Error of Mean 6.69

3. Secondary Outcome: Number and Percentage of Participants With Improved Performance (>= 30 m) in the Six Minute Walk Test (6MWT) - FAS
Description: The proportion of patients with improved performance (>= 30 meters) in the six-minute walk test (6MWT) was assessed by treatment group.
Time Frame: Baseline, Week 12
Population: The Full Analysis Set (FAS) was considered.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 302 | 302
Participants
  No | 142 | 153
  Yes | 149 | 129
  Missing | 11 | 20
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; FAS population; Test type: Other; Odds Ratio (OR) = 1.228, 95% CI 2-sided [0.882 to 1.708]

4. Secondary Outcome: Number and Percentage of Participants With Improved Performance (>= 30 m) in the Six Minute Walk Test (6MWT) - FAS Subset Without AE/SAE
Description: as for outcome 3
Time Frame: Baseline, Week 12
Population: The Full Analysis Set (FAS) population subset without AE/SAE was considered.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 290 | 294
Participants
  No | 133 | 146
  Yes | 149 | 129
  Missing | 8 | 19
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; FAS subset without AE/SAE; Test type: Other; Odds Ratio (OR) = 1.251, 95% CI 2-sided [0.895 to 1.748]

5. Secondary Outcome: Number and Percentage of Participants With Improved Performance (>= 30 m) in the 6MWT Which Walked Equal to or Less Than 300 Meters at Baseline - FAS
Description: The proportion of patients with improved performance (>= 30 meters) in the six-minute walk test (6MWT) was assessed by treatment group in a subset of patients with baseline six-minute walk distance equal to or less than 300 meters.
Time Frame: Baseline, Week 12
Population: The Full Analysis Set (FAS) was considered for patients with Baseline 6MWT equal to or less than 300 meters.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 78 | 65
Participants
  No | 35 | 31
  Yes | 41 | 29
  Missing | 2 | 5
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; FAS population; Test type: Other; Odds Ratio (OR) = 1.250, 95% CI 2-sided [0.634 to 2.464]

6. Secondary Outcome: Number and Percentage of Participants With Improved Performance (>= 30 m) in the 6MWT Which Walked Equal to or Less Than 300 Meters at Baseline - FAS Subset Without AE/SAE
Description: as for outcome 5
Time Frame: Baseline, Week 12
Population: The Full Analysis Set (FAS) population subset without AE/SAE was considered for patients with Baseline 6MWT equal to or less than 300 meters.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 75 | 63
Participants
  No | 33 | 30
  Yes | 41 | 29
  Missing | 1 | 4
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; FAS subset without AE/SAE; Test type: Other; Odds Ratio (OR) = 1.280, 95% CI 2-sided [0.644 to 2.544]

7. Secondary Outcome: Number and Percentage of Participants With Improved Performance (>= 30 m) in the 6MWT Which Walked 100-450 Meters at Baseline - FAS
Description: The proportion of patients with improved performance (>= 30 meters) in the six-minute walk test (6MWT) was assessed by treatment group in a subset of patients with baseline six-minute walk distance from 100 to 450 meters.
Time Frame: Baseline, Week 12
Population: The Full Analysis Set (FAS) was considered for patients with Baseline 6MWT between 100 or above and less than 450 meters.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 238 | 238
Participants
  No | 109 | 121
  Yes | 122 | 105
  Missing | 7 | 12
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; FAS population; Test type: Other; Odds Ratio (OR) = 1.250, 95% CI 2-sided [0.863 to 1.811]

8. Secondary Outcome: Number and Percentage of Participants With Improved Performance (>= 30 m) in the 6MWT Which Walked 100-450 Meters at Baseline - FAS Subset Without AE/SAE
Description: as for outcome 7
Time Frame: Baseline, Week 12
Population: The Full Analysis Set (FAS) population subset without AE/SAE was considered for patients with Baseline 6MWT between 100 or above and less than 450 meters.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 230 | 231
Participants
  No | 103 | 115
  Yes | 122 | 105
  Missing | 5 | 11
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; FAS subset without AE/SAE; Test type: Other; Odds Ratio (OR) = 1.260, 95% CI 2-sided [0.865 to 1.834]

9. Secondary Outcome: Change From Baseline (Week 0) in the Six Minute Walk Test (6MWT) at Weeks 4 and 8
Description: The impact of LCZ696 (Sacubitril/Valsartan) and Enalapril on functional exercise capacity was measured by the Six Minute Walk Test at Weeks 4 and 8. The 6MWT measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is able to self-pace and rest as needed as they traverse back and forth along a marked walkway.
Time Frame: Baseline, Week 4 and Week 8
Population: The Full Analysis Set (FAS) and FAS population subset without AE/SAE were considered.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 302 | 302
meters
  Baseline (FAS): number analyzed (Participants) | 301 | 300
  Baseline (FAS) | 365.37 (108.18) | 371.08 (104.41)
  Week 4 (FAS): number analyzed (Participants) | 295 | 289
  Week 4 (FAS) | 385.22 (110.55) | 385.02 (109.92)
  Change from BL at Week 4 (FAS): number analyzed (Participants) | 295 | 287
  Change from BL at Week 4 (FAS) | 19.13 (49.16) | 13.72 (51.39)
  Week 8 (FAS): number analyzed (Participants) | 291 | 284
  Week 8 (FAS) | 395.28 (112.05) | 391.72 (108.99)
  Change from BL at Week 8 (FAS): number analyzed (Participants) | 290 | 282
  Change from BL at Week 8 (FAS) | 28.72 (57.99) | 21.15 (52.75)
  Baseline (FAS without AE/SAE): number analyzed (Participants) | 289 | 292
  Baseline (FAS without AE/SAE) | 364.72 (106.86) | 371.18 (105.13)
  Week 4 (FAS without AE/SAE): number analyzed (Participants) | 284 | 283
  Week 4 (FAS without AE/SAE) | 384.58 (107.69) | 385.92 (110.81)
  Change from BL at Week 4 (FAS without AE/SAE): number analyzed (Participants) | 284 | 281
  Change from BL at Week 4 (FAS without AE/SAE) | 18.91 (49.63) | 14.45 (51.48)
  Week 8 (FAS without AE/SAE): number analyzed (Participants) | 280 | 278
  Week 8 (FAS without AE/SAE) | 396.64 (110.65) | 391.82 (109.72)
  Change from BL at Week 8 (FAS without AE/SAE): number analyzed (Participants) | 279 | 276
  Change from BL at Week 8 (FAS without AE/SAE) | 30.38 (57.07) | 21.51 (52.99)
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 4 (FAS); Test type: Other; p = 0.1814, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 4 (FAS without AE/SAE); Test type: Other; p = 0.3315, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 8 (FAS); Test type: Other; p = 0.2414, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 8 (FAS without AE/SAE); Test type: Other; p = 0.1793, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Number and Percentage of Participants Who Show Increased Levels (>= 10% Increase) of Non Sedentary Daytime Physical Activity at Week 12 Compared to Baseline
Description: Non-sedentary physical activity is defined as >= 178.50 activity counts per minute; the average number of minutes per day spent in non-sedentary physical activity will be calculated over 14 days before randomization (baseline) and the last 14 days of treatment (i.e week 10 to week 12)
Time Frame: Baseline, Week 12
Population: The Full Analysis Set was considered
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 302 | 302
Participants
  No | 175 | 163
  Yes | 28 | 31
  Missing | 99 | 108
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Increased levels (>= 10% increase) of non sedentary daytime physical activity at Week 12; Test type: Other; Odds Ratio (OR) = 0.821, 95% CI 2-sided [0.462 to 1.457]

11. Secondary Outcome: Number and Percentage of Participants Achieving PGA Score at Weeks 4, 8 and 12
Description: The Patient Global Assessment (PGA) is a self-reported tool to assess the patients' subjective rating of their disease activity widely used in HF research. The patients are asked to report functioning or response to an intervention by rating their current condition compared to their pre-intervention condition on a numerical scale: 1) much improved 2) moderately improved 3) a little improved 4) unchanged 5) a little worse 6) moderately worse or 7) much worse.
Time Frame: Week 4, Week 8, Week 12
Population: The Full Analysis Set was considered
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 302 | 302
Participants
  Week 4: Has much improved | 19 | 16
  Week 4: Has (moderately) improved | 63 | 51
  Week 4: Has a little improved | 94 | 64
  Week 4: Is unchanged | 98 | 131
  Week 4: Is a little worse | 13 | 15
  Week 4: Is (moderately) worse | 3 | 5
  Week 4: Is much worse | 1 | 1
  Week 4: Missing | 11 | 19
  Week 8: Has much improved | 23 | 24
  Week 8: Has (moderately) improved | 79 | 73
  Week 8: Has a little improved | 88 | 82
  Week 8: Is unchanged | 82 | 88
  Week 8: Is a little worse | 14 | 11
  Week 8: Is (moderately) worse | 2 | 3
  Week 8: Is much worse | 0 | 1
  Week 8: Missing | 14 | 20
  Week 12: Has much improved | 35 | 40
  Week 12: Has (moderately) improved | 72 | 67
  Week 12: Has a little improved | 82 | 74
  Week 12: Is unchanged | 79 | 94
  Week 12: Is a little worse | 12 | 7
  Week 12: Is (moderately) worse | 5 | 3
  Week 12: Is much worse | 2 | 2
  Week 12: Missing | 15 | 15
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Week 4; Test type: Other; p = 0.0516, Chi-squared
Statistical Analysis 2: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Week 8; Test type: Other; p = 0.9025, Chi-squared
Statistical Analysis 3: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Week 12; Test type: Other; p = 0.6713, Chi-squared

12. Secondary Outcome: Number and Percentage of Participants With Improved Symptoms of Heart Failure as Assessed by Patient Global Assessment (PGA)
Description: The Patient Global Assessment (PGA) is a self-reported tool to assess the patients' subjective rating of their disease activity widely used in HF research. The patients are asked to report functioning or response to an intervention by rating their current condition compared to their pre-intervention condition on a numerical scale: 1) much improved 2) moderately improved 3) a little improved 4) unchanged 5) a little worse 6) moderately worse or 7) much worse. Patients with improved symptoms were categorized as: Improvement, Is unchanged, Gets worse or Missing.
Time Frame: Week 4, Week 8, Week 12
Population: The Full Analysis Set was considered
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 302 | 302
Participants
  Week 4: Improvement | 176 | 131
  Week 4: Is unchanged | 98 | 131
  Week 4: Gets worse | 17 | 21
  Week 4: Missing | 11 | 19
  Week 8: Improvement | 190 | 179
  Week 8: Is unchanged | 82 | 88
  Week 8: Gets worse | 16 | 15
  Week 8: Missing | 14 | 20
  Week 12: Improvement | 189 | 181
  Week 12: Is unchanged | 79 | 94
  Week 12: Gets worse | 19 | 12
  Week 12: Missing | 15 | 15
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Week 4; Test type: Other; p = 0.0029, Chi-squared
Statistical Analysis 2: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Week 8; Test type: Other; p = 0.7754, Chi-squared
Statistical Analysis 3: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Week 12; Test type: Other; p = 0.2172, Chi-squared

13. Secondary Outcome: Change From Baseline in Mean Daily Non-sedentary Daytime Activity in Weekly Intervals
Description: Non-sedentary physical activity is defined as >= 178.50 activity counts per minute; Mean daily non-sedentary daytime physical activity were being calculated over weekly and compared to before the inclusion.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11 and Week 12
Population: The Full Analysis Set was considered
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 302 | 302
minutes
  Baseline: number analyzed (Participants) | 259 | 257
  Baseline | 512.07 (126.37) | 505.31 (129.74)
  Week 1: number analyzed (Participants) | 290 | 292
  Week 1 | 527.34 (129.54) | 509.28 (131.75)
  Change from BL at Week 1: number analyzed (Participants) | 250 | 250
  Change from BL at Week 1 | 22.60 (62.33) | 9.88 (50.17)
  Week 2: number analyzed (Participants) | 285 | 292
  Week 2 | 531.19 (133.89) | 508.70 (133.69)
  Change from BL at Week 2: number analyzed (Participants) | 247 | 250
  Change from BL at Week 2 | 22.80 (70.25) | 6.19 (55.14)
  Week 3: number analyzed (Participants) | 275 | 282
  Week 3 | 525.98 (126.66) | 513.63 (130.58)
  Change from BL at Week 3: number analyzed (Participants) | 238 | 241
  Change from BL at Week 3 | 13.55 (66.74) | 6.40 (62.63)
  Week 4: number analyzed (Participants) | 273 | 275
  Week 4 | 519.45 (133.21) | 503.25 (139.48)
  Change from BL at Week 4: number analyzed (Participants) | 236 | 234
  Change from BL at Week 4 | 11.99 (60.10) | -5.35 (72.35)
  Week 5: number analyzed (Participants) | 241 | 220
  Week 5 | 507.46 (129.31) | 501.70 (138.78)
  Change from BL at Week 5: number analyzed (Participants) | 212 | 190
  Change from BL at Week 5 | 1.77 (71.74) | -10.95 (81.39)
  Week 6: number analyzed (Participants) | 232 | 214
  Week 6 | 504.15 (131.05) | 500.39 (136.08)
  Change from BL at Week 6: number analyzed (Participants) | 205 | 185
  Change from BL at Week 6 | -0.44 (76.32) | -7.91 (69.71)
  Week 7: number analyzed (Participants) | 230 | 215
  Week 7 | 495.06 (127.80) | 503.46 (139.69)
  Change from BL at Week 7: number analyzed (Participants) | 202 | 187
  Change from BL at Week 7 | -10.35 (76.94) | -6.54 (75.77)
  Week 8: number analyzed (Participants) | 230 | 213
  Week 8 | 497.62 (130.56) | 496.45 (139.12)
  Change from BL at Week 8: number analyzed (Participants) | 202 | 186
  Change from BL at Week 8 | -9.49 (79.10) | -9.21 (75.23)
  Week 9: number analyzed (Participants) | 235 | 222
  Week 9 | 496.74 (128.90) | 497.24 (131.02)
  Change from BL at Week 9: number analyzed (Participants) | 205 | 196
  Change from BL at Week 9 | -10.09 (69.93) | -10.75 (75.82)
  Week 10: number analyzed (Participants) | 239 | 219
  Week 10 | 495.53 (130.97) | 500.88 (138.35)
  Change from BL at Week 10: number analyzed (Participants) | 207 | 194
  Change from BL at Week 10 | -9.46 (80.47) | -7.52 (77.12)
  Week 11: number analyzed (Participants) | 232 | 214
  Week 11 | 492.28 (127.19) | 495.14 (135.54)
  Change from BL at Week 11: number analyzed (Participants) | 201 | 192
  Change from BL at Week 11 | -12.93 (74.12) | -11.64 (75.35)
  Week 12: number analyzed (Participants) | 232 | 214
  Week 12 | 492.28 (127.19) | 495.14 (135.54)
  Change from BL at Week 12: number analyzed (Participants) | 201 | 192
  Change from BL at Week 12 | -12.93 (74.12) | -11.64 (75.35)
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 1; Test type: Other; p = 0.0008, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 2; Test type: Other; p = 0.0008, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 3; Test type: Other; p = 0.0297, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 4; Test type: Other; p = 0.0069, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 5; Test type: Other; p = 0.2275, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 6; Test type: Other; p = 0.3486, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 7; Test type: Other; p = 0.6800, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 8; Test type: Other; p = 0.7184, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 9; Test type: Other; p = 0.5301, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 10; Test type: Other; p = 0.6019, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 11; Test type: Other; p = 0.8229, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 12; Test type: Other; p = 0.8229, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Change From Baseline in Mean Daily Non-sedentary Daytime Activity in Two-weekly Intervals
Description: Non-sedentary physical activity is defined as >= 178.50 activity counts per minute; Mean daily non-sedentary daytime physical activity were being calculated over two-weekly intervals and compared to before the inclusion.
Time Frame: Baseline, Weeks 0 to 2, Weeks 2 to 4, Weeks 4 to 6, Weeks 6 to 8, Weeks 8 to 10, Weeks 10 to 12
Population: The Full Analysis Set was considered
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 302 | 302
minutes
  Baseline: number analyzed (Participants) | 259 | 257
  Baseline | 512.07 (126.37) | 505.31 (129.74)
  Weeks 0 to 2: number analyzed (Participants) | 286 | 292
  Weeks 0 to 2 | 529.63 (129.31) | 509.02 (129.97)
  Change from BL at Week 2: number analyzed (Participants) | 248 | 250
  Change from BL at Week 2 | 22.88 (60.90) | 8.06 (45.65)
  Weeks 2 to 4: number analyzed (Participants) | 275 | 279
  Weeks 2 to 4 | 522.30 (126.68) | 508.57 (131.41)
  Change from BL at Week 4: number analyzed (Participants) | 238 | 238
  Change from BL at Week 4 | 12.04 (54.84) | 0.55 (60.23)
  Weeks 4 to 6: number analyzed (Participants) | 236 | 216
  Weeks 4 to 6 | 505.54 (127.40) | 500.49 (135.70)
  Change from BL at Week 6: number analyzed (Participants) | 206 | 186
  Change from BL at Week 6 | 0.21 (68.47) | -10.86 (72.76)
  Weeks 6 to 8: number analyzed (Participants) | 231 | 213
  Weeks 6 to 8 | 495.94 (124.78) | 500.92 (135.26)
  Change from BL at Week 8: number analyzed (Participants) | 203 | 186
  Change from BL at Week 8 | -10.11 (71.75) | -7.62 (69.96)
  Weeks 8 to 10: number analyzed (Participants) | 240 | 221
  Weeks 8 to 10 | 496.57 (126.68) | 497.02 (132.96)
  Change from BL at Week 10: number analyzed (Participants) | 209 | 195
  Change from BL at Week 10 | -8.44 (68.35) | -8.75 (71.50)
  Weeks 10 to 12: number analyzed (Participants) | 226 | 210
  Weeks 10 to 12 | 483.20 (121.43) | 493.41 (130.00)
  Change from BL at Week 12: number analyzed (Participants) | 196 | 188
  Change from BL at Week 12 | -21.17 (68.77) | -13.93 (72.85)
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 2; Test type: Other; p = 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 4; Test type: Other; p = 0.0123, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 6; Test type: Other; p = 0.2560, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 8; Test type: Other; p = 0.5865, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 10; Test type: Other; p = 0.5463, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 12; Test type: Other; p = 0.3212, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Change From Baseline in Mean Daily Light Non-sedentary Daytime Physical Activity
Description: The average number of minutes per day spent in light non-sedentary physical activity was being calculated over 7 day epochs. Non-sedentary physical activity is defined as >= 178.5 activity counts per minute and light physical activity is defined as 178.5 - 565.5 counts per minute.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11 and Week 12
Population: The Full Analysis Set was considered
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 302 | 302
minutes
  Baseline: number analyzed (Participants) | 259 | 257
  Baseline | 251.94 (50.54) | 247.30 (58.70)
  Week 1: number analyzed (Participants) | 290 | 292
  Week 1 | 263.17 (55.85) | 251.37 (58.13)
  Change from BL at Week 1: number analyzed (Participants) | 250 | 250
  Change from BL at Week 1 | 14.10 (31.15) | 6.28 (27.98)
  Week 2: number analyzed (Participants) | 285 | 292
  Week 2 | 262.42 (55.12) | 248.33 (57.81)
  Change from BL at Week 2: number analyzed (Participants) | 247 | 250
  Change from BL at Week 2 | 10.91 (36.10) | 1.58 (28.80)
  Week 3: number analyzed (Participants) | 275 | 282
  Week 3 | 261.80 (52.68) | 251.12 (57.48)
  Change from BL at Week 3: number analyzed (Participants) | 238 | 241
  Change from BL at Week 3 | 9.68 (33.10) | 3.61 (31.85)
  Week 4: number analyzed (Participants) | 273 | 275
  Week 4 | 256.10 (52.61) | 246.97 (58.06)
  Change from BL at Week 4: number analyzed (Participants) | 236 | 234
  Change from BL at Week 4 | 5.14 (31.12) | -1.77 (33.49)
  Week 5: number analyzed (Participants) | 241 | 220
  Week 5 | 253.98 (54.75) | 243.71 (59.17)
  Change from BL at Week 5: number analyzed (Participants) | 212 | 190
  Change from BL at Week 5 | 2.71 (37.90) | -5.77 (37.14)
  Week 6: number analyzed (Participants) | 232 | 214
  Week 6 | 252.10 (56.73) | 244.25 (57.33)
  Change from BL at Week 6: number analyzed (Participants) | 205 | 185
  Change from BL at Week 6 | 1.08 (38.80) | -4.72 (36.44)
  Week 7: number analyzed (Participants) | 230 | 215
  Week 7 | 251.02 (52.09) | 244.85 (57.32)
  Change from BL at Week 7: number analyzed (Participants) | 202 | 187
  Change from BL at Week 7 | -0.88 (38.88) | -3.18 (37.27)
  Week 8: number analyzed (Participants) | 230 | 213
  Week 8 | 251.46 (52.21) | 245.02 (59.31)
  Change from BL at Week 8: number analyzed (Participants) | 202 | 186
  Change from BL at Week 8 | -1.71 (38.69) | -2.41 (36.53)
  Week 9: number analyzed (Participants) | 235 | 222
  Week 9 | 250.04 (52.64) | 254.84 (56.31)
  Change from BL at Week 9: number analyzed (Participants) | 205 | 196
  Change from BL at Week 9 | -2.54 (35.74) | -4.52 (37.14)
  Week 10: number analyzed (Participants) | 239 | 219
  Week 10 | 248.33 (54.44) | 245.62 (58.69)
  Change from BL at Week 10: number analyzed (Participants) | 207 | 194
  Change from BL at Week 10 | -3.43 (42.11) | -2.65 (36.76)
  Week 11: number analyzed (Participants) | 232 | 214
  Week 11 | 248.19 (53.09) | 244.83 (59.77)
  Change from BL at Week 11: number analyzed (Participants) | 201 | 192
  Change from BL at Week 11 | -3.86 (39.67) | -3.13 (34.23)
  Week 12: number analyzed (Participants) | 183 | 173
  Week 12 | 239.30 (52.76) | 243.63 (56.92)
  Change from BL at Week 12: number analyzed (Participants) | 161 | 157
  Change from BL at Week 12 | -11.98 (42.07) | -6.55 (35.79)
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 1; Test type: Other; p = 0.0004, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 2; Test type: Other; p = 0.0009, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 3; Test type: Other; p = 0.0094, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 4; Test type: Other; p = 0.0301, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 5; Test type: Other; p = 0.1557, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 6; Test type: Other; p = 0.6461, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 7; Test type: Other; p = 0.9759, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 8; Test type: Other; p = 0.3941, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 9; Test type: Other; p = 0.7209, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 10; Test type: Other; p = 0.4444, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 11; Test type: Other; p = 0.7247, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 12; Test type: Other; p = 0.2933, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Change From Baseline in Mean Daily Moderate-to-Vigorous Non-sedentary Daytime Physical Activity
Description: The average number of minutes per day spent in moderate to vigorous non-sedentary physical activity was being calculated over 7 day epochs. Non-sedentary physical activity is defined as >= 178.5 activity counts per minute and moderate-to-vigorous activity is defined as > 565.5 counts per minute.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11 and Week 12
Population: The Full Analysis Set was considered
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 302 | 302
minutes
  Baseline: number analyzed (Participants) | 259 | 257
  Baseline | 260.13 (110.94) | 258.01 (111.73)
  Week 1: number analyzed (Participants) | 290 | 292
  Week 1 | 264.16 (109.31) | 257.92 (111.47)
  Change from BL at Week 1: number analyzed (Participants) | 250 | 250
  Change from BL at Week 1 | 8.50 (45.86) | 3.60 (39.79)
  Week 2: number analyzed (Participants) | 285 | 292
  Week 2 | 268.77 (114.83) | 260.37 (116.00)
  Change from BL at Week 2: number analyzed (Participants) | 247 | 250
  Change from BL at Week 2 | 11.89 (50.98) | 4.61 (45.53)
  Week 3: number analyzed (Participants) | 275 | 282
  Week 3 | 264.19 (108.10) | 262.51 (111.15)
  Change from BL at Week 3: number analyzed (Participants) | 238 | 241
  Change from BL at Week 3 | 3.87 (49.53) | 2.80 (51.23)
  Week 4: number analyzed (Participants) | 273 | 275
  Week 4 | 263.35 (114.86) | 256.28 (115.82)
  Change from BL at Week 4: number analyzed (Participants) | 236 | 234
  Change from BL at Week 4 | 6.85 (43.45) | -3.58 (56.76)
  Week 5: number analyzed (Participants) | 241 | 220
  Week 5 | 253.48 (108.52) | 257.99 (115.65)
  Change from BL at Week 5: number analyzed (Participants) | 212 | 190
  Change from BL at Week 5 | -0.93 (51.57) | -5.18 (66.01)
  Week 6: number analyzed (Participants) | 232 | 214
  Week 6 | 252.05 (108.75) | 256.14 (115.35)
  Change from BL at Week 6: number analyzed (Participants) | 205 | 185
  Change from BL at Week 6 | -1.52 (55.23) | -3.19 (54.72)
  Week 7: number analyzed (Participants) | 230 | 215
  Week 7 | 244.04 (105.32) | 258.61 (118.51)
  Change from BL at Week 7: number analyzed (Participants) | 202 | 187
  Change from BL at Week 7 | -9.47 (57.67) | -3.35 (56.28)
  Week 8: number analyzed (Participants) | 230 | 213
  Week 8 | 246.16 (109.03) | 251.42 (113.84)
  Change from BL at Week 8: number analyzed (Participants) | 202 | 186
  Change from BL at Week 8 | -7.78 (57.13) | -6.80 (57.90)
  Week 9: number analyzed (Participants) | 235 | 222
  Week 9 | 246.70 (106.78) | 251.40 (108.51)
  Change from BL at Week 9: number analyzed (Participants) | 205 | 196
  Change from BL at Week 9 | -7.55 (54.98) | -6.23 (57.68)
  Week 10: number analyzed (Participants) | 239 | 219
  Week 10 | 247.20 (107.41) | 255.26 (116.88)
  Change from BL at Week 10: number analyzed (Participants) | 207 | 194
  Change from BL at Week 10 | -6.03 (57.08) | -4.86 (59.50)
  Week 11: number analyzed (Participants) | 232 | 214
  Week 11 | 244.09 (104.33) | 250.31 (113.81)
  Change from BL at Week 11: number analyzed (Participants) | 201 | 192
  Change from BL at Week 11 | -9.07 (51.95) | -8.51 (61.45)
  Week 12: number analyzed (Participants) | 183 | 173
  Week 12 | 237.15 (100.32) | 248.08 (113.51)
  Change from BL at Week 12: number analyzed (Participants) | 161 | 157
  Change from BL at Week 12 | -20.52 (58.37) | -11.57 (64.90)
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 1; Test type: Other; p = 0.0854, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 2; Test type: Other; p = 0.0528, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 3; Test type: Other; p = 0.4137, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 4; Test type: Other; p = 0.0082, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 5; Test type: Other; p = 0.7908, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 6; Test type: Other; p = 0.6499, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 7; Test type: Other; p = 0.5547, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 8; Test type: Other; p = 0.6961, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 9; Test type: Other; p = 0.5946, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 10; Test type: Other; p = 0.8957, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 11; Test type: Other; p = 0.8468, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 12; Test type: Other; p = 0.1711, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Total Weekly Time Spent in Non-sedentary Daytime Physical Activity
Description: Non-sedentary physical activity is defined as >= 178.5 activity counts per minute; The total time spent in non-sedentary physical activity was being calculated for each patient in weekly intervals and the temporal course for each patient was assessed.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11 and Week 12
Population: The Full Analysis Set was considered
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 302 | 302
minutes
  Baseline: number analyzed (Participants) | 264 | 263
  Baseline | 3616.87 (964.92) | 3528.56 (993.10)
  Week 1: number analyzed (Participants) | 290 | 292
  Week 1 | 3676.46 (923.85) | 3560.10 (916.16)
  Change from BL at Week 1: number analyzed (Participants) | 255 | 256
  Change from BL at Week 1 | 103.29 (509.20) | 82.48 (588.19)
  Week 2: number analyzed (Participants) | 285 | 292
  Week 2 | 3691.24 (953.03) | 3557.71 (940.60)
  Change from BL at Week 2: number analyzed (Participants) | 251 | 256
  Change from BL at Week 2 | 76.23 (563.79) | 52.38 (600.08)
  Week 3: number analyzed (Participants) | 275 | 282
  Week 3 | 3668.25 (894.91) | 3580.54 (922.70)
  Change from BL at Week 3: number analyzed (Participants) | 242 | 246
  Change from BL at Week 3 | 25.28 (571.36) | 34.56 (663.68)
  Week 4: number analyzed (Participants) | 273 | 275
  Week 4 | 3608.39 (936.87) | 3482.15 (991.15)
  Change from BL at Week 4: number analyzed (Participants) | 240 | 239
  Change from BL at Week 4 | 5.10 (497.55) | -56.23 (748.35)
  Week 5: number analyzed (Participants) | 241 | 220
  Week 5 | 3488.43 (944.87) | 3458.65 (973.75)
  Change from BL at Week 5: number analyzed (Participants) | 214 | 196
  Change from BL at Week 5 | -116.74 (607.31) | -79.18 (817.71)
  Week 6: number analyzed (Participants) | 232 | 214
  Week 6 | 3519.12 (922.58) | 3489.15 (962.55)
  Change from BL at Week 6: number analyzed (Participants) | 207 | 191
  Change from BL at Week 6 | -72.08 (569.61) | -21.73 (724.96)
  Week 7: number analyzed (Participants) | 230 | 215
  Week 7 | 3444.52 (892.15) | 3502.67 (977.43)
  Change from BL at Week 7: number analyzed (Participants) | 205 | 192
  Change from BL at Week 7 | -143.38 (605.25) | -36.18 (709.43)
  Week 8: number analyzed (Participants) | 230 | 213
  Week 8 | 3466.82 (936.51) | 3457.74 (993.56)
  Change from BL at Week 8: number analyzed (Participants) | 205 | 190
  Change from BL at Week 8 | -130.59 (631.30) | -59.92 (716.74)
  Week 9: number analyzed (Participants) | 235 | 222
  Week 9 | 3470.69 (913.06) | 3447.28 (932.67)
  Change from BL at Week 9: number analyzed (Participants) | 208 | 199
  Change from BL at Week 9 | -131.28 (549.54) | -108.48 (719.58)
  Week 10: number analyzed (Participants) | 239 | 219
  Week 10 | 3444.77 (947.18) | 3489.68 (964.08)
  Change from BL at Week 10: number analyzed (Participants) | 212 | 197
  Change from BL at Week 10 | -119.41 (648.17) | -68.93 (711.22)
  Week 11: number analyzed (Participants) | 232 | 214
  Week 11 | 3406.56 (910.84) | 3436.96 (971.78)
  Change from BL at Week 11: number analyzed (Participants) | 205 | 194
  Change from BL at Week 11 | -170.14 (632.53) | -120.35 (707.11)
  Week 12: number analyzed (Participants) | 183 | 173
  Week 12 | 3093.96 (913.14) | 3234.90 (991.50)
  Change from BL at Week 12: number analyzed (Participants) | 165 | 158
  Change from BL at Week 12 | -506.82 (792.71) | -339.15 (786.06)
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 1; Test type: Other; p = 0.0065, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 2; Test type: Other; p = 0.0316, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 3; Test type: Other; p = 0.1342, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 4; Test type: Other; p = 0.0252, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 5; Test type: Other; p = 0.9024, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 6; Test type: Other; p = 0.9052, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 7; Test type: Other; p = 0.2870, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 8; Test type: Other; p = 0.3174, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 9; Test type: Other; p = 0.5020, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 10; Test type: Other; p = 0.4037, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 11; Test type: Other; p = 0.4823, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 12; Test type: Other; p = 0.1090, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Total Weekly Time Spent in Light Non-sedentary Daytime Physical Activity
Description: Light non-sedentary daytime physical activity is defined as between 178.5 - 565.5 counts per minute; The time spent in light non-sedentary physical activity was being calculated for each patient in weekly intervals and the temporal course for each patient was assessed.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11 and Week 12
Population: The Full Analysis Set was considered
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 302 | 302
minutes
  Baseline: number analyzed (Participants) | 264 | 263
  Baseline | 1773.14 (392.22) | 1721.50 (452.26)
  Week 1: number analyzed (Participants) | 290 | 292
  Week 1 | 1834.71 (400.46) | 1757.76 (407.14)
  Change from BL at Week 1: number analyzed (Participants) | 255 | 256
  Change from BL at Week 1 | 81.84 (255.91) | 53.74 (282.22)
  Week 2: number analyzed (Participants) | 285 | 292
  Week 2 | 1823.86 (396.55) | 1736.64 (407.45)
  Change from BL at Week 2: number analyzed (Participants) | 251 | 256
  Change from BL at Week 2 | 46.26 (301.74) | 17.26 (280.12)
  Week 3: number analyzed (Participants) | 275 | 282
  Week 3 | 1826.38 (376.72) | 1751.95 (410.11)
  Change from BL at Week 3: number analyzed (Participants) | 242 | 246
  Change from BL at Week 3 | 46.05 (281.11) | 24.88 (313.52)
  Week 4: number analyzed (Participants) | 273 | 275
  Week 4 | 1778.88 (372.86) | 1707.68 (410.73)
  Change from BL at Week 4: number analyzed (Participants) | 240 | 239
  Change from BL at Week 4 | 9.17 (275.92) | -18.74 (346.02)
  Week 5: number analyzed (Participants) | 241 | 220
  Week 5 | 1745.87 (406.21) | 1683.08 (429.50)
  Change from BL at Week 5: number analyzed (Participants) | 214 | 196
  Change from BL at Week 5 | -36.66 (307.01) | -37.98 (369.53)
  Week 6: number analyzed (Participants) | 232 | 214
  Week 6 | 1759.09 (397.67) | 1701.89 (405.01)
  Change from BL at Week 6: number analyzed (Participants) | 207 | 191
  Change from BL at Week 6 | -17.85 (290.75) | -16.56 (343.51)
  Week 7: number analyzed (Participants) | 230 | 215
  Week 7 | 1747.03 (366.43) | 1702.58 (399.11)
  Change from BL at Week 7: number analyzed (Participants) | 205 | 192
  Change from BL at Week 7 | -32.03 (307.16) | -17.71 (322.33)
  Week 8: number analyzed (Participants) | 230 | 213
  Week 8 | 1750.02 (377.35) | 1705.09 (424.99)
  Change from BL at Week 8: number analyzed (Participants) | 205 | 190
  Change from BL at Week 8 | -37.50 (323.19) | -17.49 (318.83)
  Week 9: number analyzed (Participants) | 235 | 222
  Week 9 | 1746.73 (375.07) | 1706.26 (407.89)
  Change from BL at Week 9: number analyzed (Participants) | 208 | 199
  Change from BL at Week 9 | -36.47 (289.67) | -43.21 (341.30)
  Week 10: number analyzed (Participants) | 239 | 219
  Week 10 | 1724.72 (395.95) | 1712.55 (412.82)
  Change from BL at Week 10: number analyzed (Participants) | 212 | 197
  Change from BL at Week 10 | -46.95 (339.81) | -22.01 (314.65)
  Week 11: number analyzed (Participants) | 232 | 214
  Week 11 | 1717.08 (386.33) | 1697.81 (429.44)
  Change from BL at Week 11: number analyzed (Participants) | 205 | 194
  Change from BL at Week 11 | -60.08 (319.85) | -40.52 (313.76)
  Week 12: number analyzed (Participants) | 183 | 173
  Week 12 | 1559.62 (428.02) | 1607.33 (449.83)
  Change from BL at Week 12: number analyzed (Participants) | 165 | 158
  Change from BL at Week 12 | -210.49 (390.17) | -144.96 (339.29)
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 1; Test type: Other; p = 0.0061, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 2; Test type: Other; p = 0.0143, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 3; Test type: Other; p = 0.0708, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 4; Test type: Other; p = 0.0750, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 5; Test type: Other; p = 0.8017, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 6; Test type: Other; p = 0.7956, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 7; Test type: Other; p = 0.3499, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 8; Test type: Other; p = 0.1192, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 9; Test type: Other; p = 0.5237, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 10; Test type: Other; p = 0.3902, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 11; Test type: Other; p = 0.4228, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 12; Test type: Other; p = 0.1571, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Total Weekly Time Spent in Moderate-to-Vigorous Non-sedentary Daytime Physical Activity
Description: Moderate-to-vigorous non-sedentary physical activity is defined as > 565.5 counts per minute. The total time spent in moderate-to-vigorous non-sedentary physical activity was being calculated for each patient in weekly intervals and the temporal course for each patient was assessed.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11 and Week 12
Population: The Full Analysis Set was considered
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 302 | 302
minutes
  Baseline: number analyzed (Participants) | 264 | 263
  Baseline | 1843.73 (830.30) | 1807.07 (815.89)
  Week 1: number analyzed (Participants) | 290 | 292
  Week 1 | 1841.76 (769.54) | 1802.34 (775.36)
  Change from BL at Week 1: number analyzed (Participants) | 255 | 256
  Change from BL at Week 1 | 21.45 (373.16) | 28.75 (404.20)
  Week 2: number analyzed (Participants) | 285 | 292
  Week 2 | 1867.37 (806.56) | 1821.07 (813.27)
  Change from BL at Week 2: number analyzed (Participants) | 251 | 256
  Change from BL at Week 2 | 29.97 (383.31) | 35.13 (432.43)
  Week 3: number analyzed (Participants) | 275 | 282
  Week 3 | 1841.87 (755.88) | 1828.59 (777.65)
  Change from BL at Week 3: number analyzed (Participants) | 242 | 246
  Change from BL at Week 3 | -20.77 (425.19) | 9.68 (458.99)
  Week 4: number analyzed (Participants) | 273 | 275
  Week 4 | 1829.51 (801.93) | 1774.46 (815.93)
  Change from BL at Week 4: number analyzed (Participants) | 240 | 239
  Change from BL at Week 4 | -4.07 (344.29) | -37.49 (506.27)
  Week 5: number analyzed (Participants) | 241 | 220
  Week 5 | 1742.56 (767.53) | 1775.57 (798.92)
  Change from BL at Week 5: number analyzed (Participants) | 214 | 196
  Change from BL at Week 5 | -80.08 (423.07) | -41.20 (577.49)
  Week 6: number analyzed (Participants) | 232 | 214
  Week 6 | 1760.03 (763.64) | 1787.26 (810.30)
  Change from BL at Week 6: number analyzed (Participants) | 207 | 191
  Change from BL at Week 6 | -54.23 (416.05) | -5.17 (509.74)
  Week 7: number analyzed (Participants) | 230 | 215
  Week 7 | 1697.49 (732.18) | 1800.09 (829.37)
  Change from BL at Week 7: number analyzed (Participants) | 205 | 192
  Change from BL at Week 7 | -111.35 (438.85) | -18.47 (505.11)
  Week 8: number analyzed (Participants) | 230 | 213
  Week 8 | 1716.80 (769.31) | 1752.65 (802.46)
  Change from BL at Week 8: number analyzed (Participants) | 205 | 190
  Change from BL at Week 8 | -93.09 (429.65) | -42.43 (522.80)
  Week 9: number analyzed (Participants) | 235 | 222
  Week 9 | 1723.96 (750.60) | 1741.02 (757.26)
  Change from BL at Week 9: number analyzed (Participants) | 208 | 199
  Change from BL at Week 9 | -94.81 (407.63) | -65.27 (492.38)
  Week 10: number analyzed (Participants) | 239 | 219
  Week 10 | 1720.06 (760.72) | 1777.14 (811.27)
  Change from BL at Week 10: number analyzed (Participants) | 212 | 197
  Change from BL at Week 10 | -72.46 (442.80) | -46.92 (514.49)
  Week 11: number analyzed (Participants) | 232 | 214
  Week 11 | 1689.48 (731.77) | 1739.15 (803.36)
  Change from BL at Week 11: number analyzed (Participants) | 205 | 194
  Change from BL at Week 11 | -110.06 (432.47) | -79.83 (516.05)
  Week 12: number analyzed (Participants) | 183 | 173
  Week 12 | 1534.35 (678.12) | 1627.57 (778.70)
  Change from BL at Week 12: number analyzed (Participants) | 165 | 158
  Change from BL at Week 12 | -296.33 (525.81) | -194.19 (564.53)
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 1; Test type: Other; p = 0.3231, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 2; Test type: Other; p = 0.3519, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 3; Test type: Other; p = 0.8335, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 4; Test type: Other; p = 0.0465, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 5; Test type: Other; p = 0.5016, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 6; Test type: Other; p = 0.5941, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 7; Test type: Other; p = 0.2019, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 8; Test type: Other; p = 0.4125, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 9; Test type: Other; p = 0.5702, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 10; Test type: Other; p = 0.4752, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 11; Test type: Other; p = 0.5343, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 12; Test type: Other; p = 0.0985, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Change From Baseline in Peak Six Minutes of Daytime Physical Activity
Description: The peak 6 min walk (M6min) is a parameter derived by validated algorithms of the software that are used to preprocess actigraphy data. The parameter reflected the peak 6 minutes of day time physical activity. The mean daily 6-minute walking test was being calculated over 14 day intervals.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8 and Week 12
Population: The Full Analysis Set was considered
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
Number analyzed (Participants) | 302 | 302
minutes
  Baseline: number analyzed (Participants) | 259 | 257
  Baseline | 189.08 (67.75) | 182.52 (60.09)
  Week 2: number analyzed (Participants) | 285 | 292
  Week 2 | 193.54 (77.30) | 184.46 (59.49)
  Change from BL at Week 2: number analyzed (Participants) | 247 | 250
  Change from BL at Week 2 | 6.18 (46.72) | 3.52 (32.16)
  Week 4: number analyzed (Participants) | 273 | 275
  Week 4 | 191.86 (80.21) | 181.11 (61.75)
  Change from BL at Week 4: number analyzed (Participants) | 236 | 234
  Change from BL at Week 4 | 5.47 (50.93) | -0.23 (40.44)
  Week 6: number analyzed (Participants) | 232 | 214
  Week 6 | 191.21 (77.38) | 181.11 (55.07)
  Change from BL at Week 6: number analyzed (Participants) | 205 | 185
  Change from BL at Week 6 | 2.69 (42.51) | -1.02 (38.82)
  Week 8: number analyzed (Participants) | 230 | 213
  Week 8 | 183.96 (70.54) | 180.92 (57.28)
  Change from BL at Week 8: number analyzed (Participants) | 202 | 186
  Change from BL at Week 8 | -2.71 (41.43) | -0.22 (38.05)
  Week 12: number analyzed (Participants) | 183 | 173
  Week 12 | 184.42 (67.09) | 180.44 (55.36)
  Change from BL at Week 12: number analyzed (Participants) | 161 | 157
  Change from BL at Week 12 | -1.07 (49.32) | -2.45 (39.15)
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 2; Test type: Other; p = 0.4525, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 4; Test type: Other; p = 0.0445, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 6; Test type: Other; p = 0.1158, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 8; Test type: Other; p = 0.3901, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: LCZ696 (Sacubitril/Valsartan) vs Enalapril; Change from BL at Week 12; Test type: Other; p = 0.7725, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for the maximum duration of participants' treatment exposure plus any follow up period, approximately 4 months.
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Enalapril
All-Cause Mortality (participants affected / at risk) | 1/309 | 4/310
Serious Adverse Events (participants affected / at risk) | 19/309 | 28/310
Other Adverse Events (participants affected / at risk) | 168/309 | 143/310
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (Sacubitril/Valsartan) (N=309) | Enalapril (N=310)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 4 | 7
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Coronary bypass thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Stroke in evolution (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Urogenital haemorrhage (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Renal lithiasis prophylaxis (Surgical and medical procedures) | 0 | 1
Intermittent claudication (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (Sacubitril/Valsartan) (N=309) | Enalapril (N=310)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 2 | 3
Cardiac failure (Cardiac disorders) | 7 | 11
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 3 | 2
Sinus bradycardia (Cardiac disorders) | 1 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 2
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 3 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Blepharitis (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 1
Retinal vein occlusion (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 3 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Aerophagia (Gastrointestinal disorders) | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 8 | 6
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 2
Odynophagia (Gastrointestinal disorders) | 0 | 1
Rectal ulcer (Gastrointestinal disorders) | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 3
Chest discomfort (General disorders) | 1 | 1
Chest pain (General disorders) | 5 | 0
Fatigue (General disorders) | 6 | 6
Feeling abnormal (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Malaise (General disorders) | 2 | 0
Mucosal dryness (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 5 | 3
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Swelling (General disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 6 | 2
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Chlamydial infection (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 8 | 8
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 2
Rhinitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 2 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 3 | 3
Viral infection (Infections and infestations) | 3 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Drug dispensing error (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 5
Foreign body (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 2 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Underdose (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood 25-hydroxycholecalciferol decreased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 6 | 5
Blood potassium decreased (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 4 | 4
Blood pressure ambulatory decreased (Investigations) | 1 | 0
Blood pressure decreased (Investigations) | 3 | 0
Blood pressure increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Glomerular filtration rate decreased (Investigations) | 2 | 0
Glomerular filtration rate increased (Investigations) | 1 | 0
Heart rate decreased (Investigations) | 1 | 0
Heart rate increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 2 | 0
Laboratory test abnormal (Investigations) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Platelet count increased (Investigations) | 1 | 0
Red blood cell sedimentation rate increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 3 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 22 | 11
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 9
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ageusia (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 17 | 10
Dizziness postural (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 4
Hypotonia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Libido decreased (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 2 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Bladder neck obstruction (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Nocturia (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Renal disorder (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 4 | 0
Renal impairment (Renal and urinary disorders) | 4 | 3
Renal pain (Renal and urinary disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Madarosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Inguinal hernia repair (Surgical and medical procedures) | 0 | 1
Blood pressure fluctuation (Vascular disorders) | 1 | 2
Circulatory collapse (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 43 | 20
Intermittent claudication (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 3 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral coldness (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT02900378/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT02900378/SAP_001.pdf